CLINICAL TRIAL: NCT01679548
Title: Prospective Randomized Comparison of Single-port and Three-port Laparoscopic Assisted Vaginal Hysterectomy
Brief Title: Study of Laparoendoscopic Single Site Hysterectomy in Benign and Preinvasive Uterine Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LESS-H
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Benign or Preinvasive Uterine Disease
Keywords: LESS; Benign uterine disease; LAVH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-port LAVH group (Experimental): single-port laparoscopic assisted vaginal hysterectomy
  Interventions: Procedure: Single-port LAVH
- Three-port LAVH group (Active Comparator): three-port laparoscopic assisted vaginal hysterectomy
  Interventions: Procedure: Three-port LAVH

INTERVENTIONS:
Procedure: Single-port LAVH — LESS LAVH was performed using a commercially available four-channel, single-port system. A rigid, 0-degree, 5 mm laparoscope was used.
  Arms: Single-port LAVH group
Procedure: Three-port LAVH — Conventional LAVH was performed using three ports; a 12, 10, and 5-mm port was placed in the umbilicus, left lower quadrant, and suprapubic area, respectively. A rigid, 0-degree, 12 mm laparoscope was introduced through 12mm port of umbilicus.
  Arms: Three-port LAVH group

SUMMARY:
To compare the efficacy between single-port and three-port laparoscopic assisted vaginal hysterectomy in patients with benign or preinvasive uterine disease

DETAILED DESCRIPTION:
This study intended to conduct a randomized trial to determine whether LESS LAVH has a faster recovery rate than three-port LAVH.

ELIGIBILITY:
Inclusion Criteria:

* Patient who undergo laparoscopic assisted vaginal hysterectomy due to following gynecologic disease

  1. uterine leiomyoma
  2. uterine adenomyosis
  3. Endometrial hyperplasia
  4. cervical intraepithelial neoplasia including carcinoma in situ
  5. Dysfunctional uterine bleeding
  6. Other benign gynecologic disease requiring hysterectomy
* American Society of Anesthesiologists Physical Status classification I-II
* Patient who have signed an written informed consent

Exclusion Criteria:

* Uncontrolled medical disease
* Active infectious disease
* Previous pelvic radiation therapy
* Patient who requiring further procedure excluding hysterectomy, unilateral or bilateral salpingooophorectomy / salpingectomy / oophorectomy
* Patient who undergoes subtotal hysterectomy
* Patient who have other pain source excluding gynecologic disease
* Pregnancy and lactating woman

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2012-11-23 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
postoperative hospital stay | within 1 week after surgery
  The primary endpoint was to compare average length of postoperative hospital stay and the ratio of patients discharged within 2 days after surgery between LESS and conventional groups.

SECONDARY OUTCOMES:
postoperative pain | within 1 week after surgery
  Postoperative pain was recorded using the Visual Analog Pain Scale (VAS), scored from 1 to 10 (0 is no pain and 10 is agonizing pain)
postoperative analgesics requirement | within 1 week after surgery
  Whenever patients requested additional analgesia, they were administered parenterally.
operating time | 1 day (immediately ater surgery)
  skin to skin operation time was recorded
Transfusion requirement and amount | within 1 week after surgery
  Transfusion requirement and amount were recorede
intra and postoperative complication | within 1 months after surgery
  intra and post operative complications were recorede

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hyun Nam, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang OJ, Nam JH, Park JY. Comparison of single-site and three-port hysterectomy for benign uterine diseases: A randomised trial (LESS-H). Eur J Obstet Gynecol Reprod Biol. 2025 Apr 17;308:251-256. doi: 10.1016/j.ejogrb.2025.03.005. Epub 2025 Mar 10. PMID 40088545